CLINICAL TRIAL: NCT02783963
Title: Optical Coherence Tomography in Patients With Acute Myocardial Infarction and Nonobstructive Coronary Artery Disease: OCT and CMR Study (SOFT-MI)
Brief Title: Optical Coherence Tomography in Patients With Acute Myocardial Infarction and Nonobstructive Coronary Artery Disease
Acronym: SOFT-MI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Cardiology, Warsaw, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IP2014 034073
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Myocardial Infarction
Keywords: Coronary Artery Disease; Coronary Thrombosis; Coronary Stenosis; Tomography, Optical Coherence; Magnetic Resonance Imaging
MeSH Terms: conditions — Myocardial Infarction; Coronary Artery Disease; Coronary Thrombosis; Coronary Stenosis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MI with nonobstructive CAD at coronary angiography (Other): MI with nonobstructive CAD investigated by means of OCT and CMR
  Interventions: Device: OCT and CMR imaging

INTERVENTIONS:
Device: OCT and CMR imaging — OCT: Imaging for the presence and vulnerability of coronary plaque as well as plaque disruption.
  CMR: Imaging for identification of myocardial injury (late gadolinium enhancement and myocardial edema) as well as other concomitant findings.

SUMMARY:
The purpose of this study is to evaluate the prevalence and morphological features of coronary plaques by means of OCT in patients with acute myocardial infarction but without any significant coronary stenosis at coronary angiography. In addition, cardiac magnetic resonance imaging (CMR) will be performed to assess the prevalence, location, and pattern of myocardial injury as well as other concomitant findings. As a secondary analysis, the association between the distribution and characteristics of coronary plaques detected on OCT and myocardial injury shown by CMR will be evaluated. In addition, a post-hoc survey regarding the potential modification of the interventional treatment approach based on OCT analysis will be conducted.

DETAILED DESCRIPTION:
The mechanism of myocardial infarction in patients with nonobstructive coronary artery disease remains unknown. The SOFT-MI study has been designed as a single-center, prospective observational trial to investigate the prevalence of vulnerable and disrupted plaques in patients with acute MI but without any significant coronary stenosis (defined as stenosis of >50%) at coronary angiography. All patients will undergo coronary OCT immediately after coronary angiography. In addition, CMR will be performed within 1 week of coronary angiography to evaluate associated myocardial abnormalities as well as extracardiac findings. The study will provide insight into the mechanism of MI without obstructive coronary artery disease at coronary angiography, and may be useful in order to establish an appropriate therapeutic strategy for the secondary prevention of ischemic events.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of myocardial infarction: elevation of troponin to above the laboratory upper limit of normal (ULN) or new ST segment elevation of ≥1mm on 2 contiguous ECG leads or new left bundle branch block
* Symptoms of ischaemia (chest pain or anginal equivalent symptoms at rest or new onset exertional anginal equivalent symptoms with concomitant ST-segment depression, T wave inversion or transient ST-segment elevation)
* Delivery of an informed consent and compliance with study protocol
* Age ≥ 18 years

Exclusion Criteria:

* Prior diagnosis of obstructive CAD (including history of percutaneous coronary intervention or coronary artery bypass grafting)
* Stenosis >50% of any coronary vessel on invasive angiography
* Contraindication to OCT in the opinion of the treating physician
* Use of vasospastic agents
* Alternate causes of myocardial injury/ischaemia (severe anaemia, hypertensive crisis, acute heart failure, cardiac trauma, pulmonary embolism, etc.)
* Severe renal failure (eGFR<30)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-04; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Prevalence of plaque disruption | 1 day
  Prevalence of plaque disruption (including plaque rupture, plaque erosion, intracoronary thrombus) in OCT
Prevalence of myocardial injury | 1 week
  Prevalence of late gadolinium enhancement and myocardial edema in CMR

SECONDARY OUTCOMES:
Prevalence of plaque vulnerability | 1 day
  Prevalence of plaque vulnerability (including thin-cap fibroatheroma, superficial microcalcification, macrophage infiltration, and microchannel formation) in OCT
Correlation of OCT plaque characteristics and CMR findings | 1 week
Impact of OCT analysis on modification of interventional cardiology approach as well as medical treatment compared with coronary angiography alone (post-hoc analysis) | 1 week
Quantification of CAD in coronary angiography | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Maksymilian P. Opolski, MD, PhD, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (1):
- Institute of Cardiology, Warsaw, Poland

REFERENCES:
- [Derived] Opolski MP, Spiewak M, Marczak M, Debski A, Knaapen P, Schumacher SP, Staruch AD, Grodecki K, Chmielak Z, Lazarczyk H, Kukula K, Tyczynski P, Pregowski J, Dabrowski M, Kadziela J, Florczak E, Skrobisz A, Witkowski A. Mechanisms of Myocardial Infarction in Patients With Nonobstructive Coronary Artery Disease: Results From the Optical Coherence Tomography Study. JACC Cardiovasc Imaging. 2019 Nov;12(11 Pt 1):2210-2221. doi: 10.1016/j.jcmg.2018.08.022. Epub 2018 Oct 17. PMID 30343070